CLINICAL TRIAL: NCT00233974
Title: Axillary Lymph Nodes and PET (Positron Emission Tomography) Probe-Guided Surgical Resection in Locally Advanced Breast Cancer Patients: Molecular Marker Profile and Response to Neoadjuvant Chemotherapy
Brief Title: Molecular Marker Profiling of Axillary Lymph Nodes in Predicting Response in Patients With Locally Advanced or Metastatic Breast Cancer Who Are Undergoing Chemotherapy Followed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 9924; CDR0000439444 (Other: PDQ number)
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PET negative (Experimental): Traditional breast Surgery and full axillary dissection
  Interventions: Procedure: PET (positron emission tomography)
- PET positive (Experimental): PET-probe-guided breast resection and full axillary dissection
  Interventions: Procedure: PET (positron emission tomography)

INTERVENTIONS:
Procedure: PET (positron emission tomography) — Following conventional segmental mastectomy with or without needle localization, the patient will then undergo intraoperative PET-probe evaluation

SUMMARY:
RATIONALE: Comparing results of diagnostic procedures, such as molecular marker profiling, done before and after chemotherapy, may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase II trial is studying how well molecular marker profiling of axillary lymph nodes works in predicting response in patients with locally advanced or metastatic breast cancer who are undergoing chemotherapy followed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether molecular markers in pretreatment axillary lymph node metastases can predict pathologic response to neoadjuvant chemotherapy in patients with locally advanced or early metastatic breast cancer.

Secondary

* Compare molecular markers in axillary lymph node metastases with those in the primary breast tumor (obtained in protocol UNC-LCCC-9819) in patients treated with neoadjuvant chemotherapy.
* Determine changes in molecular markers in lymph nodes before and after treatment with neoadjuvant chemotherapy in these patients.
* Determine the proportion of clinical axillary lymph node-negative patients who have histopathologically node-positive disease identified by sentinel lymph node biopsy.
* Determine the rate of breast preservation in patients with large breast cancers treated with neoadjuvant chemotherapy followed by fludeoxyglucose F 18 positron emission tomography probe-guided surgical resection.

OUTLINE: Patients undergo open surgical biopsy of axillary lymph nodes OR intraoperative lymphatic mapping and sentinel lymphadenectomy for clinically node-positive or clinically node-negative disease, respectively, before and after neoadjuvant chemotherapy. The axillary lymph node tissue is examined for molecular and protein markers by immunohistochemistry and fluorescence in situ hybridization. Patients also undergo fludeoxyglucose F 18 positron emission tomography (FDG-PET) once before and then once after neoadjuvant chemotherapy. Beginning 1 hour before surgery, patients receive an injection of FDG and then undergo conventional segmental mastectomy (lumpectomy) with or without needle localization followed by FDG-PET probe-guided surgical resection of any remaining FDG-avid tumor tissue.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer by fine needle aspiration or biopsy

  * Locally advanced or early metastatic disease
* Clinically or radiographically measurable disease
* Planning to receive neoadjuvant chemotherapy for locally advanced or early metastatic disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Not specified

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for this malignancy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-05; Primary Completion 2005-02 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Improved breast conservation rates in neoadjuvant patients | 12 weeks
  Determine if an intraoperative positron emission tomography (PET) probe can improve breast conservation rates in patients treated initially with neoadjuvant chemotherapy by at least 2%.

CONTACTS AND LOCATIONS:
Overall Officials: David W. Ollila, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States